CLINICAL TRIAL: NCT03067740
Title: Intraperitoneal Dexmedetomidine as an Adjuvant to Bupivacaine for Management of Pain in Children Undergoing Laparoscopic Appendicectomy: A Prospective Randomized Trial
Brief Title: Intraperitoneal Dexmedetomidine for Post-laparoscopic Appendicectomy Pain Management in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ali Elnabtity, Principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: approved on 11 june 2016
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Pain, Postoperative
Keywords: appendicectomy; children; local anesthetics; laparoscopy; peritoneum
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine group (Active Comparator): intraperitoneal instillation of bupivacaine 0.25% ( 2mg/kg) after excision of the appendix.
  Interventions: Drug: Bupivacaine
- Bupivacaine-Dexmedetomidine group (Experimental): intraperitoneal instillation of bupivacaine 0.25% ( 2mg/kg) plus dexmedetomidine 1mcg/kg after excision of the appendix.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — intraperitoneal instillation of bupivacaine 0.25% ( 2mg/kg) after excision of the appendix.
  Other Names: Marcaine
  Arms: Bupivacaine group
Drug: Dexmedetomidine — intraperitoneal instillation of bupivacaine 0.25% ( 2mg/kg) plus dexmedetomidine 1mcg/kg after excision of the appendix.
  Other Names: Precidex
  Arms: Bupivacaine-Dexmedetomidine group

SUMMARY:
Fifty two children of American Society of Anesthesiologists (ASA) physical status I and II, aged 8-14 years old, of both gender, with suspected acute appendicitis scheduled for laparoscopic appendicectomy, were included in this study. Patients were randomized into group (B) and group (BD) with a 1:1 allocation ratio.At the end of surgery, and after peritoneal lavage, those patients who were allocated to B group (bupivacaine group; n = 26) received bupivacaine 0.25% intraperitoneally at a dose of 2 mg/kg followed by 5 ml normal saline. However, in group BD (bupivacaine, Dexmedetomidine group; n = 26), bupivacaine 0.25% at a dose of 2mg/kg was instilled intraperitoneally followed by dexmedetomidine 1mcg/kg diluted in 5 ml normal saline. In the postoperative period, assessments were made for pain and sedation on awakening in PACU (0 time) and at 2, 4, 6, 12,and 24 h. Abdominal and/or shoulder pain was assessed on the 10-cm Visual Analog Scale (VAS). Sedation was assessed using the Ramsay sedation score. Also the occurrence of nausea or vomiting was recorded . The time from extubation to the first administration of pethidine was registered. The consumption of postoperative analgesia was recorded. Side effects of the study drugs were assessed and recorded by the ward nurses for 24h postoperatively. Possible complications such as respiratory depression, allergic reactions, local anaesthetic toxicity,dizziness, , headache, were recorded and managed accordingly. Duration of surgery and length of stay in PACU were noted. Before discharge to home, length of stay in the hospital was recorded and parent's satisfaction was assessed using the 7-point Likert scale

DETAILED DESCRIPTION:
A written informed consent for participation in the trial was obtained by parents or the legal guardians . Fifty two children participate in the study.

Randomization and blindness: Patients were randomized into group (B) and group (BD) with a 1:1 allocation ratio. The allocated intervention was written on a slip of paper, placed in a sealed serially numbered, opaque envelopes. The envelopes were serially opened, and the allocated intervention was implemented. Patients were equally distributed in both groups. All investigators, parents, and patients were blind to which method was being used.

Study description:

On arrival to the operating room, routine preoperative evaluation was performed, and the procedure was explained to all parents. Before premedication, patients and parents were instructed in the use of the 10-cm Visual Analog Scale (VAS),with score raging from 0 (no pain) to 10 (worst pain imaginable). Baseline measurements of heart rate (HR), mean arterial pressure (MAP), respiratory rate (RR), and room air oxygen saturation (SaO2) were obtained using an electrocardiogram, a "Dinamap" automated blood pressure monitor, and a pulse oximeter, respectively.

All children received premedication with midazolam 0.05 mg/kg intravenously afterward, Ringer's lactate infusion (20 ml/kg/h) was started. Standardized prophylactic antiemetic was iv ondansetron 0.15 mg/kg. General anesthesia was inducted with propofol 2 mg/kg, rocuronium 0.6 mg/kg, and fentanyl 2 mcg/kg intravenously (i.v.). Endotracheal intubation was performed, tube size was calculated according to the formula: age/4+4. Anesthesia was maintained with a sevoflurane and oxygen mixture, with total fresh gas flow 3 L/min controlled by mechanical ventilation, tidal volume 5-10 ml/kg. The respiratory rate adjusted according to the end tidal CO2 (maintaining CO2 in the normal range of 35-45 mmHg). Standardized prophylactic antiemetic was ondansetron 0.15 mg/kg.

In both study groups, laparoscopic surgery was performed according to the standard surgical protocol. Local infiltration of port sites was performed by 4 ml xylocaine 1% at a maximum dose of 3 mg/kg. Standardized surgery involved 3 ports, a 5 or10-mm umbilical Hasson cannula and 3 or 5- mm left iliac fossa and suprapubic ports. Pneumoperitoneum was achieved using nonhumidified and nonheated CO2, with the intra-abdominal pressure maintained around 10-12 mmHg.

At the end of surgery, and after peritoneal lavage, those patients who were allocated to B group (bupivacaine group; n = 26) received bupivacaine 0.25% intraperitoneally at a dose of 2 mg/kg followed by 5 ml normal saline. However, in group BD (bupivacaine, Dexmedetomidine group; n = 26), bupivacaine 0.25% at a dose of 2mg/kg was instilled intraperitoneally followed by dexmedetomidine 1mcg/kg diluted in 5 ml normal saline. Surgeons instilled the study solution through a suction-irrigation device under visual control onto the parietal and visceral peritoneum of the right iliac fossa and pelvis to cover the appendix stump, lower pole of the cecum, and the terminal ileum. At the end of the operation, CO2 was cleared completely from the peritoneal cavity by manual compression of the abdomen with open trocar. Patients in both groups received intravenous paracetamol 15 mg/kg (Perfalgan, Bristol-Myers Squibb Pharmaceuticals Ltd, New York City, NY, USA).

Reversal of the muscle relaxant was carried out using prostigmine at a dose of 0.05-0.07 mg/kg and atropine at a dose of 0.02 mg/kg. The patients were then transferred to the postanaesthesia care unit (PACU) where monitoring of heart rate (HR), mean arterial blood pressure (MAP), respiratory rate (RR), arterial oxygen saturation (SaO2), and pain scoring was carried out. After operation, paracetamol 15mg/kg iv drip was administered on a regular base every 8h, and iv pethidine 1mg/kg as rescue analgesia ( whenVAS≥ 4) for the 1st 24. the occurrence of nausea or vomiting was recorded and patients were immediately given ondansetron 0.15 mg/kg if they experienced nausea and/or vomiting.

The ward nurses were instructed to omit the 6-h dose of pethidine if they considered that the patient was over sedated or pain free.

The time from extubation to the first administration of pethidine was registered. Side effects of the study drugs were assessed and recorded by the ward nurses for 24h postoperatively. Oxygen desaturation was considered when SpO2 dropped below 93% for more than 10 s. Bradycardia was defined as a HR 20% decrease from the baseline, whereas a HR more than 20% of the baseline was labeled as tachycardia. A drop in MAP by 20% or more of the baseline was regarded as hypotension while a MAP value higher than the baseline by 20% was regarded as hypertension. Other possible complications such as respiratory depression, allergic reactions, local anaesthetic toxicity,dizziness, , headache, were recorded and managed accordingly.

The primary outcome of the study:

In the postoperative period, assessments were made for pain on awakening in PACU (0 time) and at 2, 4, 6, 12,and 24 h. Abdominal and/or shoulder pain was assessed on the 10-cm Visual Analog Scale (VAS).

The secondary outcomes of the study:

* Sedation scores at PACU time and at 2h, 4h, 6h, 12h, and 24h after surgery.
* Time of first request of analgesia.
* Amount of rescue pethidine in 24h after surgery.
* Duration of surgery.
* Length of stay in PACU.
* Frequency of nausea and vomiting and other complications after surgery.
* Length of stay in hospital after surgery.
* Parents satisfaction before discharge to home.

Sample size calculation:

To calculate the sample size, the postoperative opioid consumption at day 1 in a similar clinical setting was taken into account. With a 2-tailed α = 0.05 and a power of 80%, we needed 23 patients in each group. Considering the anticipated drop out as 10%, 52 patients were asked to participate in the study. Data will be presented as a mean ± standard deviation, median, numbers, and frequencies, as appropriate. Statistical significance accepted at a P < 0.05 Statistical analysis will be performed using SPSS program version 19 (Armonk, NY: IBM Corp.) and EP16 program. Student's t-test, Chi-square test, Mann-Whitney U-test, and Fisher's exact test will be used for statistical analysis, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients are of American Society of Anesthesiologists (ASA) physical status I and II, aged 8-14 years old, of both gender, with suspected acute appendicitis scheduled for laparoscopic appendicectomy.

Exclusion Criteria:

* The diagnosis of developmental delay, attention deficit disorder, chronic pain, psychiatric illness, previous open abdominal surgery, the presence of a gastrostomy, ventricular-peritoneal shunt or other abdominal prosthesis, immunosuppression, and those allergic to any of the medications.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative abdominal and/or shoulder VAS pain score | at the start of postanesthesia care unit (PACU)(0 time), and 2 Hours, 4 Hours, 6 Hours, 12 Hours, and 24 Hours postoperative
  assessment of changes in pain scores along different time intervals in the postoperative 24 hours

SECONDARY OUTCOMES:
Time of first request of analgesia. | from the start of postanesthesia care unit (PACU time) and up to 8 hours
  when VAS becomes more than 3, analgesia is given and the time is recorded
amount of rescue pethidine consumed | in 24 Hours postoperative
  in milligrams
Length of hospital stay | from end of surgery till discharge to home, up to one week
  postoperative stay in hospital (days)
Sedation score | at the start of postanesthesia care unit (PACU)(0 time), and 2 Hours, 4 Hours, 6 Hours, 12 Hours, and 24 Hours postoperative
  Ramsay Sedation Score (RSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Elnabtity, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witt WP, Weiss AJ, Elixhauser A. Overview of Hospital Stays for Children in the United States, 2012. 2014 Dec. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #187. Available from http://www.ncbi.nlm.nih.gov/books/NBK274247/ PMID 25695124
- [Result] Sauerland S, Lefering R, Neugebauer EA. Laparoscopic versus open surgery for suspected appendicitis. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD001546. doi: 10.1002/14651858.CD001546.pub2. PMID 15495014
- [Result] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060
- [Result] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Result] El-Labban GM, Hokkam EN, El-Labban MA, Morsy K, Saadl S, Heissam KS. Intraincisional vs intraperitoneal infiltration of local anaesthetic for controlling early post-laparoscopic cholecystectomy pain. J Minim Access Surg. 2011 Jul;7(3):173-7. doi: 10.4103/0972-9941.83508. PMID 22022099
- [Result] Golubovic S, Golubovic V, Cindric-Stancin M, Tokmadzic VS. Intraperitoneal analgesia for laparoscopic cholecystectomy: bupivacaine versus bupivacaine with tramadol. Coll Antropol. 2009 Mar;33(1):299-302. PMID 19408641
- [Result] Albanese AM, Albanese EF, Mino JH, Gomez E, Gomez M, Zandomeni M, Merlo AB. Peritoneal surface area: measurements of 40 structures covered by peritoneum: correlation between total peritoneal surface area and the surface calculated by formulas. Surg Radiol Anat. 2009 Jun;31(5):369-77. doi: 10.1007/s00276-008-0456-9. Epub 2009 Jan 14. PMID 19142561
- [Result] Kahokehr A, Sammour T, Soop M, Hill AG. Intraperitoneal use of local anesthetic in laparoscopic cholecystectomy: systematic review and metaanalysis of randomized controlled trials. J Hepatobiliary Pancreat Sci. 2010 Sep;17(5):637-56. doi: 10.1007/s00534-010-0271-7. PMID 20393755